CLINICAL TRIAL: NCT00570401
Title: A Phase 2 Trial of Dasatinib in Patients With Lung Adenocarcinoma With Acquired Resistance to Erlotinib or Gefitinib
Brief Title: Dasatinib in Treating Patients With Advanced Lung Cancer That Is No Longer Responding to Erlotinib or Gefitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mskcc 06-143; P30CA008748 (NIH); MSKCC-06143; BMS-MSKCC-06143; NCT00590057 (obsolete NCT alias)
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Dasatinib

ARMS (1):
- Dasatinib (Experimental): Beginning 1 week after completion of erlotinib hydrochloride or gefitinib therapy, patients receive oral dasatinib twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Response is assessed by CT scan at 4 weeks, 8 weeks, and then every 8 weeks thereafter.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well dasatinib works in treating patients with advanced lung cancer that is no longer responding to erlotinib or gefitinib.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall response rate (complete response and partial response) in patients with acquired erlotinib hydrochloride- or gefitinib-resistant advanced adenocarcinoma of the lung treated with dasatinib.

Secondary

* To determine the progression-free survival and overall survival of patients treated with this drug.
* To determine the overall response rate in patients with EGFR T790M lung adenocarcinomas treated with this drug.
* To determine the progression-free survival and overall survival of patients with EGFR T790M lung adenocarcinomas treated with this drug.
* To determine the toxicity profile of dasatinib in these patients.

OUTLINE: Beginning 1 week after completion of erlotinib hydrochloride or gefitinib therapy, patients receive oral dasatinib twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Response is assessed by CT scan at 4 weeks, 8 weeks, and then every 8 weeks thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed adenocarcinoma of the lung

  * Advanced disease
* Previously treated with erlotinib hydrochloride or gefitinib for 6 months (at any time) and meets 1 of the following criteria:

  * Previously received treatment with erlotinib hydrochloride or gefitinib* and had a radiographic partial or complete response to treatment with erlotinib hydrochloride or gefitinib as defined by RECIST or WHO criteria
  * Documented mutation in EGFR from tumor DNA NOTE: *Patients may have received other treatments subsequently including radiation or chemotherapy
* Must have developed acquired resistance to erlotinib hydrochloride or gefitinib

  * Radiographic evidence of disease progression during treatment with erlotinib hydrochloride or gefitinib
* Have previously undergone a biopsy of a site of progressive disease on protocol MSKCC 04-103* NOTE: *Results of this biopsy are not required to be enrolled on this trial
* Measurable indicator lesions have not been previously irradiated
* No CNS lesion that is symptomatic and/or requiring escalating doses of corticosteroids

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* WBC ≥ 3,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 2 mg/dL or creatinine clearance ≥ 55 mL/min
* QTc < 450 msec
* Able to take oral medications
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 weeks after study drug is stopped
* No significant medical history or unstable medical condition, including any of the following:

  * History of diagnosed congenital long QT syndrome
  * Ventricular arrhythmia
  * Congestive heart failure
  * Recent myocardial infarction
  * Unstable angina
  * Active infection
  * Uncontrolled hypertension

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior cytotoxic chemotherapy
* At least 3 weeks since prior radiation therapy to a major bone-marrow containing area
* At least 7 days since prior quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, or lidoflazine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent A. Miller, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Gregory J. Riely, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Johnson ML, Riely GJ, Rizvi NA, Azzoli CG, Kris MG, Sima CS, Ginsberg MS, Pao W, Miller VA. Phase II trial of dasatinib for patients with acquired resistance to treatment with the epidermal growth factor receptor tyrosine kinase inhibitors erlotinib or gefitinib. J Thorac Oncol. 2011 Jun;6(6):1128-31. doi: 10.1097/JTO.0b013e3182161508. PMID 21623279

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib: Dasatinib in Patients with Lung Adenocarcinoma Receiving Erlotinib with Acquired Resistance to EGFR Tyrosine Kinase Inhibitors (TKIs)
Period: Overall Study
Arm/Group | Dasatinib
Started | 21
Completed | 19
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Determine the Overall Objective Response
Description: To determine the overall response rate in patients with acquired erlotinib hydrochloride- or gefitinibresistant advanced adenocarcinoma of the lung treated with dasatinib using the RECIST criteria. Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.22 Changes in only the largest diameter (uni-dimensional measurement) of the tumor lesions are used in the RECIST.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 19
participants
  Stable Disease (SD) | 6
  Progression of Disease (POD) | 13

ADVERSE EVENTS:
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 12/21
Other Adverse Events (participants affected / at risk) | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=21)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Pleuritic pain (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=21)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (5)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
ALT, SGPT (Blood and lymphatic system disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (9)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes